CLINICAL TRIAL: NCT06619405
Title: AMD and Validating Rod-Meditated Dark Adaptation With Everyday Task Performance
Brief Title: AMD and Validation Rod-Meditated Dark Adaptation With Everyday Task Performance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Boehringer Ingelheim (Industry); StreetLab Vision (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00115500
Record Dates: First submitted 2024-09-24; First posted 2024-10-01 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Early AMD (Other): Study patients who have a diagnosis of early AMD
  Interventions: Diagnostic Test: Streetlab VR
- Intermediate AMD (Other): Study patients who have a diagnosis of Intermediate AMD
  Interventions: Diagnostic Test: Streetlab VR
- Geographic Atrophy (Other): Study patients who have a diagnosis of Geographic Atrophy
  Interventions: Diagnostic Test: Streetlab VR
- AMD Controls (Other): Study patients who have healthy eyes
  Interventions: Diagnostic Test: Streetlab VR

INTERVENTIONS:
Diagnostic Test: Streetlab VR — Streetlab VR is a virtual reality headset that is warn to simulate walking through a maze at different light levels.

SUMMARY:
The goal is to conduct a cross-sectional, single timepoint study on older adults with early and intermediate AMD, and with subretinal drusenoid deposits (SDD), and those in normal health, establishing an association between dark adaptation and reading performance under dim illumination, both which depend on rod photoreceptors.

DETAILED DESCRIPTION:
The investigators propose two sites for the study, Duke University and UAB. Each site will enroll 100 participants as indicated in the table above, per the AREDS 9-step AMD classification system, with 200 participants in the sample. Because the variance of rod-mediated dark adaptation in AMD patients increases with increasing disease severity, the investigators will implement a larger sample size for intermediate AMD and a smaller sample for patients in normal macular health.

The investigators will collect demographic characteristics (age, race/ethnicity, gender), ocular medical history from the electronic health record, and medication use. In addition, the protocol will focus on measuring the following major components:

1. Comprehensive eye exam
2. Rod-mediated dark adaptation
3. Reading performance
4. Mobility
5. Ellipsoid zone loss and attenuation

Statistical associations will be computed using correlational analysis for the overall sample, within each patient group, and also separately for those with SDD. Sample size estimation is challenging because there is no previous literature on the association between rod-mediated dark adaptation and MNREAD reading performance or MOST performance. With a sample size of 200 participants, the investigators will have adequate statistical power (80%) to detect a correlation of at least 0.20 for the total sample and adequate statistical power to detect within-group correlations of at least 0.40.

ELIGIBILITY:
Inclusion Criteria:

* Capable and willing to provide consent
* Has been diagnosed with early, intermediate dry age-related macular degeneration or geographic atrophy or has a healthy macular for controls
* At least 50 years of age

Exclusion Criteria:

* Unable or unwilling to give consent or unable to read consent since the study involves testing which requires reading
* Under 50 years of age
* Presence of dense cataracts in the study eye (s) that can affect visual function tests
* Presence of glaucoma requiring treatment during the study and/or visual field defects
* Previous retinal laser or surgical therapy in the study eye(s)
* Previous retinal laser or surgical therapy in the study eye(s)
* Any other ocular condition requiring long-term therapy or surgery during the study
* The participant has photographically significant corneal or media opacities in either eye that would preclude adequate ophthalmic imaging and functional testing
* Diagnosis of nystagmus that will interfere with testing
* High myopia -8 Diopters or more severe
* The participant has, in the opinion of the Investigator, any physical or mental condition that would increase the risk of participation in the study or may interfere with the study procedures, evaluations, and outcome assessments.

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Total number of participants with total ellipsoid zone (EZ) band attenuation | Approximately 2 years
  Total EZ attenuation is defined as EZ-RPE (retinal pigment epithelium) thickness = 0 μm.

SECONDARY OUTCOMES:
Total number of participants with partial ellipsoid zone (EZ) band attenuation | Approximately 2 years
  Partial EZ attenuation is defined as EZ-RPE (retinal pigment epithelium) thickness ≤ 20 μm.
Rod-mediated dark adaptation | Single visit, approximately 5-6 hours
  Measured for right and left eyes separately using the AdaptDx, a computerized dark adaptometer.
Reading performance as measured by the MNREAD (Minnesota low vision reading) chart | Single visit, approximately 5-6 hours
  Reading performance will be assessed binocularly with the MNREAD iPad app on a digital version of the MNREAD chart. The MNREAD is a text based chart used to measure near visual acuity in people with normal or low vision.
Mobility as measured by the Mobility Standardized Test (MOST) | Single visit, approximately 5-6 hours
  The MOST task involves walking through a maze which can be performed under a range of mesopic and photopic conditions. Scoring is automatically computed based on the duration and mobility errors, which generated a score from 0 to 100, with 100 as the best performance.

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Lad, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No